CLINICAL TRIAL: NCT00854737
Title: A Combination of Cytidine and Omega-3 Fatty Acids in Bipolar Disorder: Are There Additive or Synergistic Mood Stabilizing Effects?
Brief Title: Cytidine and Omega-3 Fatty Acids in Bipolar Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Beth L. Murphy MD, PhD, Investigator, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2009-P-000149
Record Dates: First submitted 2009-02-27; First posted 2009-03-03 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Bipolar Disorder
Keywords: bipolar disorder; bipolar depression; bipolar mania; manic depression; depression; mania; hypomania
MeSH Terms: conditions — Bipolar Disorder; Depression; Mania | interventions — Cytidine; Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Omega-3 fatty acid and cytidine supplementation
  Interventions: Dietary Supplement: cytidine; Dietary Supplement: omega-3 fatty acids
- 2 (Active Comparator): omega-3 fatty acid supplementation
  Interventions: Dietary Supplement: omega-3 fatty acids
- placebo (Placebo Comparator): placeno or sugar pill
  Interventions: Drug: placebo

INTERVENTIONS:
Dietary Supplement: cytidine — cytidine (2g po daily for 4 months)
  Arms: 1
Dietary Supplement: omega-3 fatty acids — omega-3 fatty acids (4g po daily for 4 months)
  Arms: 1; 2
Drug: placebo — sugar pill
  Other Names: arm 2 and 3
  Arms: placebo

SUMMARY:
The goal of the proposed clinical trial is to assess the effect of oral cytidine and omega-3 fatty acids (O3FA) on bipolar disorder symptoms. This study is a 4-month, randomized, parallel-group, double-blind, placebo-controlled pilot study of a combination of cytidine and omega-3 fatty acids in 90 recently ill subjects with bipolar disorder. During the 16 week period of the study, subjects are assigned to one of three groups: 1) omega-3 fatty acids + cytidine supplementation, 2) omega-3 fatty acids supplementation alone, and 3) placebo supplementation.

DETAILED DESCRIPTION:
Previous studies examining the effect of omega-3 fatty acids on bipolar depression have had mixed results. Some studies have found that omega-3 fatty acids have a positive effect on bipolar depression symptoms, while other studies have found no difference between placebo and omega-3 fatty acid treatment.

The variable effects noted with omega-3 fatty acids may be due in part to a real effect with limited potency. Larger effects might be achieved by combining agents with synergistic effects.

Cytidine is necessary to form key intermediates in the biosynthesis of the phospholipids phosphatidylcholine and phosphatidylethanolamine, which are major components of eukaryotic cell membranes. Recent human studies by our group have shown that CDP-choline (a compound composed of cytidine and choline) can modify brain phospholipid synthesis in healthy adults and may have antidepressant effects (Babb et al., 1996; Babb et al., 2002; Carlezon et al., 2002; Renshaw et al., 1999). The combination of omega-fatty acids and the related pyrimidine, uridine, was associated with enhanced antidepressant-like activity in rats (Carlezon et al., 2005). Thus, the combination of omega-3 fatty acid and cytidine, which is interconverted with uridine in the body, may provide a safe and powerful way to treat bipolar disorder, especially bipolar depression.

This study is a 4-month, randomized, parallel-group, double-blind, placebo-controlled pilot study of a combination of cytidine and omega-3 fatty acids in 90 recently ill subjects with bipolar disorder. During the 16 week period of the study, subjects are assigned to one of three groups: 1) omega-3 fatty acids + cytidine supplementation, 2) omega-3 fatty acids supplementation alone, and 3) placebo supplementation.

ELIGIBILITY:
Inclusion Criteria:

* bipolar disorder
* mood episode within past year
* stable medication regimen

Exclusion Criteria:

* primary psychiatric disorder other than bipolar disorder
* significant suicide or homicide risk
* unstable medical conditions
* current or planned pregnancy
* lactose intolerance
* medications affecting lipid absorption or metabolism
* clozapine treatment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2004-07; Primary Completion 2007-08 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Mood Rating Scale Scores | weekly-biweekly

SECONDARY OUTCOMES:
Study Retention Time | 4 months
functional recovery | weekly-biweekly

CONTACTS AND LOCATIONS:
Overall Officials: Beth L Murphy, MD, PhD, Principal Investigator — Mclean Hospital
Locations (2):
- United States (2):
  - McLean Hospital, Belmont, Massachusetts
  - Jersey Shore University Medical Center, Neptune City, New Jersey

REFERENCES:
- [Background] Babb SM, Appelmans KE, Renshaw PF, Wurtman RJ, Cohen BM. Differential effect of CDP-choline on brain cytosolic choline levels in younger and older subjects as measured by proton magnetic resonance spectroscopy. Psychopharmacology (Berl). 1996 Sep;127(2):88-94. doi: 10.1007/BF02805979. PMID 8888372
- [Background] Babb SM, Wald LL, Cohen BM, Villafuerte RA, Gruber SA, Yurgelun-Todd DA, Renshaw PF. Chronic citicoline increases phosphodiesters in the brains of healthy older subjects: an in vivo phosphorus magnetic resonance spectroscopy study. Psychopharmacology (Berl). 2002 May;161(3):248-54. doi: 10.1007/s00213-002-1045-y. Epub 2002 Mar 22. PMID 12021827
- [Background] Carlezon WA Jr, Mague SD, Parow AM, Stoll AL, Cohen BM, Renshaw PF. Antidepressant-like effects of uridine and omega-3 fatty acids are potentiated by combined treatment in rats. Biol Psychiatry. 2005 Feb 15;57(4):343-50. doi: 10.1016/j.biopsych.2004.11.038. PMID 15705349
- [Background] Stoll AL, Severus WE, Freeman MP, Rueter S, Zboyan HA, Diamond E, Cress KK, Marangell LB. Omega 3 fatty acids in bipolar disorder: a preliminary double-blind, placebo-controlled trial. Arch Gen Psychiatry. 1999 May;56(5):407-12. doi: 10.1001/archpsyc.56.5.407. PMID 10232294
- [Background] Carlezon WA, Pliakas AM, Parow AM, Detke MJ, Cohen BM, Renshaw PF. Antidepressant-like effects of cytidine in the forced swim test in rats. Biol Psychiatry. 2002 Jun 1;51(11):882-9. doi: 10.1016/s0006-3223(01)01344-0. PMID 12022961
- [Derived] Murphy BL, Stoll AL, Harris PQ, Ravichandran C, Babb SM, Carlezon WA Jr, Cohen BM. Omega-3 fatty acid treatment, with or without cytidine, fails to show therapeutic properties in bipolar disorder: a double-blind, randomized add-on clinical trial. J Clin Psychopharmacol. 2012 Oct;32(5):699-703. doi: 10.1097/JCP.0b013e318266854c. PMID 22926607
- See also: hospital website with links to research group and studies — http://www.mclean.harvard.edu